CLINICAL TRIAL: NCT01993446
Title: A Randomized, Double-blind, Vehicle Controlled Study of the Safety and Efficacy of Topical DRM02 in Subjects With Rosacea
Brief Title: A Safety and Efficacy Study of DRM02 in Subjects With Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRM02-ROS02
Record Dates: First submitted 2013-11-15; First posted 2013-11-25 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DRM02 (Experimental): DRM02 Topical Gel, 0.25%
  Interventions: Drug: DRM02
- Vehicle (Placebo Comparator): DRM02 Topical Gel, Vehicle
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: DRM02
  Arms: DRM02
Other: Vehicle
  Arms: Vehicle

SUMMARY:
The purpose of this study is to determine whether DRM02 is safe and effective in the treatment of rosacea when applied twice daily for 6 weeks.

DETAILED DESCRIPTION:
This is a double-blind, randomized, vehicle controlled, study enrolling 30 subjects with rosacea and designed to assess the safety, tolerability, and preliminary efficacy of DRM02.

Safety will be assessed during the study, through adverse events, local skin responses, urinalysis, serum chemistry and hematology laboratory testing, physical examination and vital signs.

Preliminary efficacy will be assessed through inflammatory lesion counts, the Investigator's Global Evaluation (IGE) and the Rosacea Signs and Symptoms (RSS) scale.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 70 years of age.
* Clinical diagnosis of rosacea with a score of 2 or 3 on the Investigator's Global Evaluation (IGE) of Rosacea scale and at least 15 and not more than 40 papules.
* Subjects willing to minimize external factors that might trigger rosacea flare-ups.
* Male or non-pregnant, non-lactating females.
* Signed informed consent.

Exclusion Criteria:

* Severe self-reported facial sensitivity.
* Severe sun sensitivity.
* Ocular-only, phymatous rosacea or steroid rosacea.
* Use of topical rosacea treatments in the 4 weeks prior to baseline.
* Use of systemic corticosteroids within the 4 weeks prior to baseline.
* Use of systemic antibiotics in the 4 weeks prior to baseline.
* Use of systemic retinoids for in the 6 months prior to baseline.
* Use of topical retinoids in the 3 months prior to baseline.
* Use of light- or laser-based rosacea treatments in the past 2 months prior to baseline.
* Cosmetic procedures within the 2 months prior to baseline.
* Use of topical anti-aging medications in the 2 weeks prior to baseline.
* Subjects who have poor skin condition within 5 cm of the treatment area.
* Subjects who are current drug or alcohol abusers; have a history of immunodeficiency or are a poor medical risk because of other systemic diseases or active uncontrolled infections.
* Subjects with an unstable medical condition or a medical condition not adequately controlled with standard medical therapy.
* Subjects who are actively participating in an experimental therapy study or who have received experimental therapy within 30 days.
* Subjects who have a clinically significant laboratory value at screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory lesion count | Week 6

SECONDARY OUTCOMES:
Investigator's Global Evaluation (IGE) | From baseline to weeks 0, 1, 2, 3, 4 and 6
IGE dichotomized into "success" and "failure" | Week 6
Percent change in inflammatory lesions | Week 6

OTHER OUTCOMES:
Rosacea Signs and Symptoms (RSS) | From baseline to weeks 0, 1, 2, 3, 4 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Beth Zib, Study Director — Dermira, Inc.
Locations (3):
- Canada (3):
  - Windsor Clinical Research, Inc., Windsor, Ontario
  - Clinique Médicale Dr Isabelle Delorme, Drummondville, Quebec
  - Innovaderm Research, Inc, Montreal, Quebec